CLINICAL TRIAL: NCT07395622
Title: Impact of the EpiFaith® Syringe on the Learning Curve of Anesthesia Residents for the Labor Epidural Technique: A Quasi-Experimental Study
Brief Title: EpiFaith Resident Learning Curve Trial
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Michaela Kristina Farber, MD, Chief, Division of Obstetric Anesthesiology, Mass General Brigham, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023P001926; 2023A006350 (Other Grant/Funding Number: Flat Medical)
Record Dates: First submitted 2026-01-17; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Epidural Analgesia; Epidural Analgesia for Labour and Delivery; Learning Curve
Keywords: labor epidural; learning curve; epidural syringe; anesthesia residents
MeSH Terms: interventions — Syringes

STUDY DESIGN:
Intervention Model Description: The study will be conducted as a quasi-eperimental trial. Study subjects will be assigned to one of the two groups for their epidural placement based on the month of their rotation, with alternating months: 1) EpiFaith® Group, in which EpiFaith® syringe is used; or 2) Control Group in which a conventional glass syringe is used
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control (glass epidural syringe) (Experimental)
  Interventions: Device: Control (glass) syringe
- EpiFaith syringe (Experimental)
  Interventions: Device: EpiFaith epidural syringe

INTERVENTIONS:
Device: EpiFaith epidural syringe — The EpiFaith syringe is an FDA-cleared epidural syringe.
  Arms: EpiFaith syringe
Device: Control (glass) syringe — glass epidural syringe
  Arms: Control (glass epidural syringe)

SUMMARY:
This study aims to evaluate the impact of the EpiFaith® syringe on the learning curve of anesthesia residents for the labor epidural technique. Anesthesia residents with prior experience placing < 5 labor epidurals will be enrolled. Their performance of 20 sequential labor epidural placements with either standard technique with a beveled glass syringe or the EpiFaith® syringe will be observed. Successful epidural placement over time with sequential epidural placement attempts will be measured between groups. The primary outcome will be rate of successful epidural placement. Success will be defined as a composite of 4 criteria: maximum 3 attempts for placement; no need to re-site at a different level; no required intervention by the supervising attending anesthesiologist; and adequate analgesia with a visual analog score (VAS) <3 at 30 minutes. We hypothesize that use of the EpiFaith® syringe will enable a faster learning curve for successful epidural placement. A cumulative sum chart (CUSUM) analysis will evaluate whether the EpiFaith® syringe causes deviation from the control learning curve. Secondary outcomes will include rate of inadvertent dural puncture and epidural replacement rate.

DETAILED DESCRIPTION:
The lumbar epidural technique for labor analgesia requires technical training and a manual skillset. A prior study evaluating anesthesia resident learning curves for a traditional labor epidural technique demonstrated a steep learning curve for the first 20 epidural placements, followed by a plateau with gradual proficiency maximized after 60 epidural placements (1). A prior study evaluated a spring-loaded epidural syringe among experienced providers (2). However, the impact of a spring-loaded epidural syringe on novice anesthesia resident learning curves is unknown. In addition, the impact of EpiFaith® use at the time of manual skill acquisition on success with subsequent traditional epidural technical skills is unknown.

The EpiFaith® syringe is FDA-cleared and has a spring-loaded piston designed to detect entry into the epidural space upon loss of resistance (LOR) as the epidural needle tip moves from the dense ligamentum flavum to the high-compliance epidural space. Performing the LOR technique using the EpiFaith® syringe, the piston within the syringe moves forward driven by spring force when a drop in pressure is detected. Piston movement within the syringe is visibly detectable with a yellow indicator in the syringe when LOR occurs. In a feasibility study of 40 labor epidural placements, 3 of 4 expert obstetric anesthesiology physicians reported the EpiFaith® syringe to be equal to superior in quality to the standard LOR syringe, with 100% success rate and no inadvertent dural punctures (3).

Evaluating the impact of the EpiFaith® syringe on learning curves of anesthesia residents with minimal prior technical experience will help inform how we approach education regarding the labor epidural technique. Steeper learning curves with faster time to proficiency may benefit both patients and supervising staff, while if no difference is determined, the use of the EpiFaith® syringe can be de-emphasized during the training period.

ELIGIBILITY:
Inclusion Criteria:

* Anesthesiology residents with fewer than 5 prior epidural placement experiences

Exclusion Criteria:

* anesthesiology residents with more than 5 prior epidural placement experiences

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
success of labor epidural attempt | time of epidural placement to 30 minutes after dosing of the epidural
  success of labor epidural attempt over time by each resident, with success defined as a composite requiring:
  1. Less than 3 attempts for placement
  2. No need to re-site the epidural needle
  3. No staff intervention
  4. NRS 3 or less at 30 minutes post-loading epidural dose

SECONDARY OUTCOMES:
rating of the epidural syringe | from time of placement to immediately following placement
  rating of the epidural syringe loss of resistance technique
Incidence of inadvertent dural puncture | from time of epidural placement for a maximum of 5 days
  incidence of inadvertent dural puncture
incidence of postdural puncture headache | from time of epidural placement up to 5 days
  incidence of postdural puncture headache
Need for epidural catheter replacement during labor | from time of epidural placement through delivery during hospital admission
  need for epidural catheter replacement during labor

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No